CLINICAL TRIAL: NCT02578511
Title: Standard Maintenance [POMP/D (Methotrexate, 6 - Mercaptopurine, Vincristine, Prednisone/Dexamethasone)] Plus Ixazomib Maintenance Therapy in Adults With Acute Lymphoblastic Leukemia, Lymphoblastic Lymphoma or Mixed Phenotype Acute Leukemia in Complete Remission (CR)
Brief Title: Standard Maintenance POMP/D Plus Ixazomib Maintenance Therapy in Adult Patients With Acute Lymphoblastic Leukemia, Lymphoblastic Lymphoma or Mixed Phenotype Acute Leukemia in Complete Remission (CR)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No enrollment, another competing study and difficult to find the right person to enroll on this study.
Sponsor: Ehab L Atallah (Other)
Responsible Party: Sponsor-Investigator, Ehab L Atallah, Associate Professor, Department of Medicine, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO25835
Record Dates: First submitted 2015-09-30; First posted 2015-10-19 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Acute Lymphoblastic Leukemia in Complete Remission; Lymphoblastic Lymphoma in Complete Remission; Mixed Phenotype Acute Leukemia in Complete Remission
Keywords: Acute Lymphoblastic Leukemia in Complete Remission; Lymphoblastic Lymphoma in Complete Remission; Mixed Phenotype Acute Leukemia in Complete Remission; IXAZOMIB; POMP/D; Phase I; Early Phase; Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Mixed Phenotype Acute Leukemia; ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixazomib (MLN9708) in combination with standard POMP/D (Experimental): Patients who are receiving maintenance therapy with the POMP/D (Methotrexate, 6-Mercaptopurine, Vincristine, Prednisone/Dexamethasone) will be enrolled. Each cycle will be 28 days. The patients will receive IV vincristine, dexamethasone or prednisone, methotrexate and 6 - Mercaptopurine. Ixazomib will be administered on days 1, 8 and 15.
  Both prednisone and dexamethasone are acceptable drugs in maintenance therapy. For example, in the HyperCVAD regimen or the CALGB 8811 prednisone is used. Patients will continue the same maintenance regimen they are receiving and ixazomib will be added to that.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Patients who have been on stable doses of 6 - MP, vincristine, and methotrexate for a minimum of eight weeks and have at least six months remaining of maintenance are eligible to receive Ixazomib, which will be administered on days 1, 8 and 15.

SUMMARY:
In this phase I study, escalating doses of IXAZOMIB will be combined with the POMP/D regimen.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

The primary objective is to determine the maximum-tolerated dose of IXAZOMIB (MLN9708) (maximum of 4 mg, which is the recommended phase II dose for IXAZOMIB (MLN9708) in combination with standard maintenance therapy with POMP/D (methotrexate, 6- mercaptopurine, vincristine, prednisone/dexamethasone) and to assess the tolerability of POMP/D and IXAZOMIB (MLN9708) maintenance in adult patients with acute lymphoblastic leukemia, lymphoblastic lymphoma (LBL) or mixed phenotype acute leukemia (MPAL) in complete remission (CR).

SECONDARY OBJECTIVE

To determine the three-year progression-free survival (PFS) of patients treated with oral IXAZOMIB (MLN9708) and standard maintenance regimen. Progression-free survival will be measured from the start of induction to disease relapse.

STUDY DESIGN

The maximum-tolerated dose of single agent IXAZOMIB was 1.76 to 2.0mg/m2 when given on a twice a week schedule1 and > 2.34 mg/m2 to 2.97 mg/m2 on a weekly schedule in previous studies.

Three patients will be treated per dose level unless dose-limiting toxicity (DLT) is observed. The starting dose of IXAZOMIB will be 3 mg orally on days 1, 8 and 15. If no DLT is seen in the first three patients, the dose will be increased to 4 mg on days 1, 8 and 15 in a classic 3 +3 phase I design. We will not attempt to increase the dose beyond 4 mg orally which, if achieved with acceptable toxicity, would be accepted as the recommended phase 2 dose (RP2D). Zero of three DLTs would allow escalation to the next dose level. One of three DLTs will require expanding to six patients; one of six DLTs will allow escalation again. Two DLTs will require dose de-escalation. The maximum-tolerated dose (MTD) will be the highest dose administered at which no more than one DLT was observed.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients 18 years or older.
* Have B-precursor, T cell ALL, MPAL or LBL in CR following therapy and receiving maintenance therapy. Patients with persistent minimal residual disease and/or in complete remission with incomplete platelet recovery are not eligible.
* Prior therapy: Should have achieved CR following the induction and intensification phases of treatment, with no limit on the number of prior treatment regimens, and started treatment with POMP/D maintenance. Patients who achieved CRp or CR with persistence of minimal residual disease are not eligible.
* Patients are eligible after allogeneic stem cell transplantation.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients must meet the following clinical laboratory criteria:

  * Total bilirubin < 1.5 X the upper limit of the normal range (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase. (AST) < 3 X ULN.
  * Calculated creatinine clearance > 30 mL/min.
  * Absolute neutrophil count (ANC) > 1,000/cmm and platelets > 75,000/cmm.
* Patient has a life expectancy of at least six months.
* Patients must be at least two weeks from major surgery, radiation therapy, participation in other investigational trials and have recovered from clinically significant toxicities of these prior treatments.
* Patients should be on stable doses of 6-mercaptopurine, methotrexate, vincristine and prednisone/dexamethasone as part of the POMP/D regimen, for a minimum of eight weeks PRIOR to starting ixazomib treatment.
* Patients should have at least six months of therapy with the POMP/D regimen remaining prior to starting IXAZOMIB (MLN9708).
* Female patients who:

  * Are postmenopausal for at least one year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice two effective. methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion criteria:

* Systemic treatment, within 14 days before study enrollment, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of ginkgo biloba or St. John's wort.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements. Patients should not have evidence of active infection.
* Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or GI procedure that could interfere with the oral absorption or tolerance of treatment.
* Active chronic graft vs. host disease requiring therapy.
* Patient has ≥ grade 2 peripheral neuropathy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the trial start and throughout the duration of this trial.
* Failure to have fully recovered (i.e., < grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past six months.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with treatment completion according to this protocol.
* Known allergy to any of the study medications, their analogues or excipients in the various formulations of any agent.
* Diagnosed or treated for another malignancy within two years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Female patients who are breastfeeding or have a positive serum pregnancy test during the screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of ixazomib with POMP/D maintenance | Eight (8) weeks
  The patient cohort enrolled at each dose level will be monitored for dose-limiting toxicity for eight weeks prior to enrolling the next cohort of patients at a new dose level. Subsequent patient cohorts will be enrolled at doses according to the CRM design. A maximum sample size of 12 patients will be enrolled over four potential doses to determine the maximum tolerated dose of ixazomib with POMP/D maintenance. Adverse events will be summarized with descriptive statistics at each dose level of ixazomib.

SECONDARY OUTCOMES:
Progression-free survival of patients treated with oral Ixazomib and standard maintenance regimen. | Three (3) years
  Progression-free survival will be measured from the time of diagnosis to disease relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Atallah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided